CLINICAL TRIAL: NCT07133906
Title: Accuracy of Interstitial Continuous Glucose Sensors in Neonates
Status: Not yet recruiting | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Sarbattama Rimi Sen, Vice Chair Pediatric Clinical Research, Women and Infants Hospital of Rhode Island
Other Study IDs: 2177993
Record Dates: First submitted 2025-07-22; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Hypoglycemia; Gestational Diabetes; Maternal Obesity Complicating Pregnancy; Small-for-gestational Age; Large-for-gestational Age
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal dried blood spots and cord serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pregnant women >24 weeks gestation and their infants: Pregnant women >24 weeks gestation; infants of pregnant women >24 weeks gestation, including 11 infants of women with gestational diabetes, 11 infants of women with type II diabetes, 11 infants of women with type I diabetes, 6 small-for-gestational age (SGA) infants, 6 large-for-gestational age (LGA) infants, and 12 control infants who are not considered at-risk for hypoglycemia.
  Interventions: Device: Continuous glucose monitoring; Device: Cerebral near-infrared spectroscopy

INTERVENTIONS:
Device: Continuous glucose monitoring — A blinded Abbott Freestyle Libre 3 Pro will be placed on the newborn
Device: Cerebral near-infrared spectroscopy — Blinded cerebral near infrared spectroscopy will be assessed

SUMMARY:
Low blood sugar in newborns is common and if prolonged or untreated may place them at increased risk for later learning and behavior challenges. Currently, we measure newborn glucose with at least four painful heel sticks, missing one in four episodes of low blood sugar. The goal of this observational study is to develop a less invasive approach to glucose monitoring, developed for newborns, that provides more frequent glucose measurements. We will also measure how a pregnant woman's health impacts newborn glucose, and how newborn glucose is linked to brain oxygen saturation and development.

DETAILED DESCRIPTION:
Glycemic control in newborns remains a major challenge for neonatal care. One third of U.S. infants are screened for neonatal hypoglycemia (NH) with repeated, painful heel sticks, most commonly based on dichotomous maternal diabetes determination or newborn size. Yet, less than 50% of these infants subsequently develop and are treated for hypoglycemia. If treatment is needed, it is based on "operational thresholds" that do not account for the actual effect of glycemia on brain metabolism, nor for its long-term consequences, and potentially expose infants to unnecessary treatment that may further amplify harm. Thus, both screening and treatment for NH lack precision and are not driven by physiology or outcome.

Improving NH risk stratification requires maternal metabolic and neonatal glycemic characterization in a cohort that includes dyads considered at-risk, with comparison to not-at-risk controls. Establishing "functional thresholds" for glycemic treatment requires evaluation of reliable bedside measurable proxies of brain metabolic "health" during the neonatal period. Further, these need to contextualised within the longitudinal trajectory of the domains known to be impacted by NH, namely executive and visual motor function. These critical domains have not been investigated together in one pre-birth, longitudinal cohort, and this knowledge gap has limited advancements in NH care.

* The primary objective of this observational study is to characterize the Abbott FreeStyle Libre 3 Pro continuous glucose monitoring system performance with respect to point of care whole blood reference in neonates.
* A secondary objective is to determine maternal and neonatal predictors of NH and child neurodevelopment.
* A secondary objective is to identify glycemic and cerebral saturation thresholds of exposure linked to adverse neurodevelopment.

Study Design

• Non-randomized, single arm, single-center, prospective, observational study

Study Procedures Visit 1 (V1) t: 30-36 weeks' gestation

Procedures:

* Complete the following electronic surveys and questionnaires: Demographics, Holmes-Rahe Life Stress Inventory, Infant Feeding Intentions Questionnaire, and the Fat/Sugar/Fruit/Vegetables Screener.
* Participants will be provided blood self-collection kits and asked to provide fasting blood samples at 35-37 weeks gestation, to be archived for later measurement of metabolic markers.

Visit 2 (V2): post-delivery in hospital

Procedures:

* All infants will have blinded FreeStyle Libre 3 Pro Continuous Glucose Monitors placed on the lateral thigh by the PI or trained staff which will be continued to hospital discharge or for 10 days, depending which occurs first.
* Near Infrared Spectroscopy (NIRS) probe will be placed on the forehead of the infant, connected to a monitor that will be blinded (covered) to the parents and clinical team.
* Infants will have additional research blood drawn (50 uL) by heel stick or venipuncture (based on clinical method of blood collection) at least twice.
* Any extra blood available will be used to measure ketones and lactate using a hand-held meter.
* Every effort will be made to align research blood draws with clinical draws, however, if this is not possible, enrolled infants will have an additional 1-2 heel sticks daily for research purposes.
* Infant body composition will be measured using air displacement plethysmography (PeaPod TM) and bioimpedance assay within 72 hours of life.
* Infant weight and length will be measured.
* The Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) will be administered by an NNNS trained and certified staff.
* Additional clinical data will be extracted from the both the maternal and infant medical record.

Visit 3 (V3): 6 months of life (between 5 and 7 months of age) - Parent will complete the following electronic questionnaires: 6-Month Ages and Stages Questionnaire, Breastfeeding Status Questionnaire, and the Infant Feeding Practices Survey (6 Months).

Visit 4 (V4): 1 year of life (between 11 and 13 months of age)

- Procedure: Parent will complete the following electronic questionnaires: Breastfeeding Status Questionnaire, Infant Feeding Practices Survey (12 Months), 1-Year Ages and Stages Questionnaire, Child Health Questionnaire, and the Brief Infant Toddler Social and Emotional Assessment (BITSEA).

Additional clinical data will be abstracted from the medical record of the mother and infant after discharge. Study staff will complete chart reviews for key pregnancy health variables outlined in the "Medical Record Abstraction Form" and enter into study database.

Cord blood will be collected and archived for a subset of subjects.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years or older
* speaks English, Spanish, Portuguese, or Haitian Creole
* pregnant >24 weeks gestation with singleton pregnancy

Exclusion Criteria:

* known concomitant maternal or fetal condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff
* plans to deliver at a hospital other than Women and Infants Hospital of Rhode Island

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Antenatal floor, labor and delivery unit (L&D), neonatal intensive care unit (NICU), mother baby unit (MBU), and obstetrics and diabetes clinics at Women and Infants Hospital
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Point Accuracy: System agreement analysis | From time of birth to discharge, an average of 3 days
  Number and percent of glucose monitoring (GM) sensor results within the intervals +/- 20% of glucose reference throughout the system measuring range

SECONDARY OUTCOMES:
Episodes of neonatal hypoglycemia (NH) by risk factors | Between birth to 72 hours after birth
  Count of neonatal hypoglycemia (NH) episodes in infants born with various maternal and neonatal risk factors (maternal diabetes, maternal gestational glucose intolerance, maternal obesity, fetal growth abnormalities, maternal beta blockers, and preterm delivery) or no risk factors.
NNNS scores | From time of birth to 72 hours after birth, at an average of 48 hours of age
  NNNS subscale score quartiles
ASQ scores | 6 months and 12 months
  Ages and Stages (ASQ) scores

IPD SHARING:
Plan to Share IPD: Undecided